CLINICAL TRIAL: NCT05951777
Title: Autologous Adipose-Derived Mesenchymal Stem Cells for Chronic Traumatic Brain Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Biosciences LLC (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Organization: Hope Biosciences Research Foundation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBTBI02
Record Dates: First submitted 2023-06-26; First posted 2023-07-19 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury
Keywords: severe; intracranial hemorrhage; chronic; neurological injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Lymphoma, Follicular; Intracranial Hemorrhages; Bronchiolitis Obliterans Syndrome; Trauma, Nervous System | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Autologous Adipose Derived Mesenchymal Stem Cells
  Interventions: Biological: Autologous HB-adMSCs
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: Autologous HB-adMSCs — Hope Biosciences autologous adipose-derived mesenchymal stem cells
  Arms: Treatment
Drug: Normal Saline — Sterile Saline Solution 0.9%
  Arms: Placebo

SUMMARY:
The global objective of this study is to establish the safety and investigate the potential treatment effect of an intravenous infusion of HB-adMSCs (Hope Biosciences adipose-derived mesenchymal stem cells) on brain structure, neurocognitive/functional outcomes, and neuroinflammation after traumatic brain injury.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind, placebo-controlled Phase 2a study of three infusions of autologous HB-adMSCs (Hope Biosciences adipose-derived mesenchymal stem cells) (2 x 10^8 total cells per dose) administered over a 6 week period with 14 day intervals between infusions. Subjects will be monitored and assessed for infusion related toxicity for at least 1 hour after the infusion and by telephone 24hr. after each infusion. Safety assessments will be conducted at the study follow-up clinic visits 6 and 12 months, and 2 years (telephone call) after the last HB-adMSC (Hope Biosciences adipose-derived mesenchymal stem cells) infusion, or more frequently if infusion related adverse events are suspected.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18 and 55 years of age.
2. Documented functional neurological damage to the central nervous system from closed head trauma that is unlikely to improve with present standard of care approaches.
3. A Glasgow Outcome Scale-Extended (GOS-E) score >2 and ≤6.
4. Onset or diagnosis of the injury or disease process greater than 6 months and <= 20 years.
5. Ability to obtain consent from the subject or their legally authorized representative (LAR).
6. Ability to verbally communicate in English or Spanish (required for validated neurocognitive outcome testing).

Exclusion Criteria:

1. Known history of:

   1. intellectual deficiency or uncontrolled psychiatric conditions likely to invalidate our ability to assess changes in cognition or behavior, or at the discretion of the PI,
   2. recently treated infection,
   3. renal disease or altered renal function (screening eGFR < 60 mL/min/1.73m2),
   4. hepatic disease or altered liver function (screening SGPT > 150 U/L or T. Bilirubin >1.3 mg/dL),
   5. cancer,
   6. immunosuppression (screening WBC < 3, 000 cells/ml),
   7. Positive infectious disease tests including HIV, Hep. B, Hep. C., and Syphilis,
   8. chemical or ETOH dependency that in the opinion of the investigator would preclude enrollment,
   9. acute or chronic lung disease requiring significant medication/oxygen supplementation,
   10. bleeding disorders including immune-mediated heparin-induced thrombocytopenia,
   11. known sensitivity to heparin, Lovenox, and pork products,
   12. individuals with mechanical prosthetic heart valves,
   13. individuals who have received a stem cell treatment, gene or cellular therapy.
2. Normal brain CT/MRI exam.
3. History of spinal cord injury.
4. Diagnosed with a genetic or metabolic disorder related to the neurologic condition.
5. Other acute or chronic medical conditions that, in the opinion of the investigator, may increase the risks associated with study participation.
6. For women of childbearing potential, a positive pregnancy test at the screening visit or, for both women and men, unwillingness to comply with acceptable methods of birth control.
7. Concurrent participation in interventional drug or device study.
8. Inability to undergo the diagnostic tests (PET/DT-MRI) or unwilling/unable to cooperate with the diagnostic tests and outcome assessments.
9. Metal implants including baclofen pumps that would preclude DT-MRI.
10. Unwilling or unable to return for the follow-up study visits.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glucose | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical lab evaluation of level of glucose in the blood (mg/dL)
Calcium | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical lab evaluation of level of calcium in the blood (mg/dL)
  clinical lab evaluation of level of calcium in the blood (mg/dL) clinical lab evaluation of level of calcium in the blood (mg/dL)
Albumin | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical lab evaluation of level of albumin in the blood (g/dL)
Total Protein | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical lab evaluation of total protein in the blood (g/dL)
Sodium | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical lab evaluation of total sodium in the blood (mmol/L)
Total carbon dioxide | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical lab evaluation of total carbon dioxide in the blood (mmol/L)
Potassium | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical lab evaluation of potassium in the blood (mmol/L)
Chloride | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical lab evaluation of chloride in the blood (mmol/L)
BUN (blood urea nitrogen) | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of blood urea nitrogen (BUN) (mg/dL)
Creatinine | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of creatinine in blood (mg/dL
Alkaline phosphatase | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of alkaline phosphatase (ALP) in blood (IU/L)
Alanine aminotransferase | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of alanine aminotransferase (ALT) in blood (IU/L)
Aspartate aminotransferase | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of aspartate aminotransferase (AST) in blood (IU/L)
Total Bilirubin | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of total bilirubin in blood (mg/dL)
White blood cell | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of white blood cells (WBC) in blood (x 10^3/uL)
Red blood cell | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of red blood cells (RBC) in blood (x 10^6/uL)
Hemoglobin | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of hemoglobin in blood (g/dL)
Hematocrit | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of hematocrit in blood (%)
Mean corpuscular volume | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of mean corpuscular volume (MCV) in blood (fL)
Mean corpuscular hemoglobin | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of mean corpuscular hemoglobin (MCH) in blood (pg)
Mean corpuscular hemoglobin concentration | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of mean corpuscular hemoglobin concentration (MCHC) in blood (g/dL)
Red cell distribution width | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of red cell distribution width (RDW) in blood (%)
Neutrophils | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of neutrophils in blood (%)
Lymphocytes | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of lymphocytes in blood (%)
Monocytes | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of monocytes in blood (%)
Eosinophils | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of eosinophils in blood (%)
Basophils | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of basophils in blood (%)
Absolute Neutrophils | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of absolute neutrophils in blood (x 10^3/uL)
Absolute lymphocytes | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of absolute lymphocytes in blood (x 10^3/uL)
Absolute monocytes | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of absolute monocytes in blood (x 10^3/uL)
Absolute eosinophils | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of absolute eosinophils in blood (x 10^3/uL)
Absolute basophils | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of absolute basophils in blood (x 10^3/uL)
Immature Granulocytes | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of immature granulocytes in blood (%)
Absolute Immature Granulocytes | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of absolute immature granulocytes in blood (x 10^3/uL)
Platelets | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of platelets in blood (x 10^3/uL)
Prothrombin Time | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of time for blood to coagulate (seconds)
INR (international normalized ratio) | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of international normalized ratio of blood coagulation (no unit)
Urine Pregnancy (if applicable) | Week 0 (Infusion 1), change from week 0 (Infusion 1) at week 2 (Infusion 2), change from week 0 (Infusion 1) at week 4 (Infusion 3), change from week 0 (Infusion 1) at 6 months post-infusion, change from week 0 (Infusion 1) at 1 year post-infusion
  clinical evaluation of human chorionic gonadotropin (hCG) in urine (positive/negative)

SECONDARY OUTCOMES:
Whole brain MRI (Magnetic resonance imaging) | Baseline, change from baseline at 6 months post-infusion
  DTI (Diffusion tensor imaging) to assess macro- and micro-structural properties
PET/DT-MRI (positron emission tomography/Diffusion tensor-Magnetic resonance imaging) | Baseline, change from baseline at 6 months post-infusion
  [11C]ER-176 (a Radioligand for 18-kDa (Translocator Protein)) tracer/label to identify brain proteins associated with neuroinflammatory response regulation
Glasgow Outcome Scale - Extended | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  Dichotomized-Glasgow Outcomes Score (GOSE) to evaluate affect, functional outcome, and neuropsychological function.
  Minimum score = 1 = dead; 2 = vegetative state; 3 = lower severe disability; 4 = upper severe disability; 5 = lower moderate disability; 6 = upper moderate disability; 7 = lower good recovery; Maximum score = 8 = upper good recovery;
  Higher scores indicate better outcome.
Disability Rating Scale | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  Rating of level of arousal, cognitive ability related to activities of daily living, and level of functioning.
Behavior Rating of Executive Functions-Adult | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  Behavior Regulation and Metacognitive Indices assess everyday executive functions
TBI (Traumatic Brain Injury) Quality of Life Questionnaires | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  TBI-QOL SF (Traumatic Brain Injury-Quality of Life Short-Form) measures physical, psychological health, cognitive, and participation outcomes:
  Cognition: minimum raw score = 10, maximum raw score = 50. A higher score represents better functioning.
  Communication/Comprehension: minimum raw score = 9, maximum raw score = 45. A higher score represents better functioning.
  Independence: minimum raw score = 8, maximum raw score = 40. A higher score represents better functioning.
  Mobility: minimum raw score = 9, maximum raw score = 45. A higher score represents better functioning.
  Satisfaction with Social Roles & Activities: minimum raw score = 10, maximum raw score = 50. A higher score represents better functioning.
  Upper Extremity Function: minimum raw score = 9, maximum raw score = 45. A higher score represents better functioning.
Brief Symptom Inventory 18 | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  Brief Symptom Inventory with 18 items contains three six-item scales for somatization, anxiety, depression, and the global Scale Global Severity Index (GSI). Each item is scored either 0 (Not at all), 1 (A little bit), 2 (Moderately), 3 (Quite a bit), 4 (Extremely), or R (Refused).
  The GSI therefore ranges between 0 (minimum) - 72 (maximum) and the three scales range between 0 (minimum) - 24 (maximum).
  Higher scores indicate worse outcome.
NIH Toolbox - Pattern Comparison Processing Speed Test | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  An assessment of processing speed. Participants are asked to quickly determine whether two stimuli are the same or not the same.
  Participants are measured based on reaction time (seconds) and accuracy.
NIH Toolbox - Dimensional Change Card Sort Test | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  An assessment of cognitive flexibility and attention. Participants are asked to match a series of bivalent test pictures (e.g., yellow balls and blue trucks) to the target pictures, first according to one dimension (e.g., color) and then, after a number of trials, according to the other dimension (e.g., shape).
  Participants are measured based on reaction time (seconds) and accuracy.
NIH Toolbox - Picture Vocabulary Test | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  An assessment of receptive vocabulary administered in a computer-adaptive test (CAT) format. Participants must choose which of four pictures best represents a word presented via audio.
  Participants are measured based on reaction time (seconds) and accuracy.
NIH Toolbox - List Sorting Working Memory Test | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  Designed to assess working memory (WM). List Sorting is a sequencing task requiring participants to sort and sequence stimuli that are presented visually and auditorily.
  Participants are measured based on accuracy.
NIH Toolbox - Flanker Inhibitory Control and Attention Test | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  An assessment of inhibitory control and attention. The participant is asked to focus on a particular stimulus while inhibiting attention to the stimuli flanking it.
  Participants are measured based on reaction time (seconds) and accuracy.
NIH Toolbox - 9-hole Pegboard Dexterity Test | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  The NIH Toolbox 9-Hole Pegboard Dexterity Test is a simple test of manual dexterity; it records the time required for the participant to accurately place and remove nine plastic pegs into a plastic pegboard. Raw scores are recorded as time in seconds that it takes the participant to complete the task with each hand (a separate score for each - Dominant vs. Non-Dominant Hand).
  Shorter time to complete the task indicates a better outcome. Longer time to complete the task indicates a worse outcome.
Rey Auditory Verbal Learning Test | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  Immediate learning and delayed recall of a word list
Verbal Fluency | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  Attentional control and verbal generativity
Wechsler Adult Intelligence Scale - IV: Processing Speed Index | Baseline, change from baseline at 6 months post-infusion, change from baseline at 1 year post-infusion
  Information processing rate on paper-pencil tasks requiring visual attention. It is composed of 10 core subtests and five supplemental subtests, with the 10 core subtests comprising the Full Scale IQ.
  There are four index scores representing major components of intelligence: Verbal Comprehension Index (VCI); Perceptual Reasoning Index (PRI); Working Memory Index (WMI); Processing Speed Index (PSI)
  Two broad scores are also generated, which can be used to summarize general intellectual abilities: Full Scale IQ (FSIQ), based on the total combined performance of the VCI, PRI, WMI, and PSI; General Ability Index (GAI), based only on the six subtests that comprise the VCI and PRI
  The range of possible WAIS-IV (Wechsler Adult Intelligence Scale - IV) full scale IQs is 45-155. The WAIS-IV computes scaled scores for each individual based exclusively on chronological age.
  Higher score indicates better outcome.
Plasma cytokines | Baseline imaging (visit #2), change from baseline at 6 months post-infusion, change from baseline 1 year post-infusion
  measure plasma cytokines via a bead-based, flow cytometric ELISA (enzyme-linked immunosorbent assay) for the cytokines
Interleukin 1-alpha | Baseline imaging (visit #2), change from baseline at 6 months post-infusion, change from baseline 1 year post-infusion
  measure IL-1α (Interleukin 1-alpha) via a bead-based, flow cytometric ELISA (enzyme-linked immunosorbent assay) for the cytokines
Interleukin 4 | Baseline imaging (visit #2), change from baseline at 6 months post-infusion, change from baseline 1 year post-infusion
  measure IL-4 (Interleukin 4) via a bead-based, flow cytometric ELISA (enzyme-linked immunosorbent assay) for the cytokines
Tumor necrosis factor alpha | Baseline imaging (visit #2), change from baseline at 6 months post-infusion, change from baseline 1 year post-infusion
  measure TNFα (Tumor necrosis factor alpha) via a bead-based, flow cytometric ELISA (enzyme-linked immunosorbent assay) for the cytokines
Interleukin 6 | Baseline imaging (visit #2), change from baseline at 6 months post-infusion, change from baseline 1 year post-infusion
  measure IL-6 via a bead-based, flow cytometric ELISA (enzyme-linked immunosorbent assay) for the cytokines
Interleukin 10 | Baseline imaging (visit #2), change from baseline at 6 months post-infusion, change from baseline 1 year post-infusion
  measure IL-10 (Interleukin 10) via a bead-based, flow cytometric ELISA (enzyme-linked immunosorbent assay) for the cytokines
Albumin | Baseline imaging (visit #2), change from baseline at 6 months post-infusion, change from baseline 1 year post-infusion
  measure concentration of albumin via BCG (bromocresol green) immunochemical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Cox, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Memorial Hermann Hospital / UTHealth McGovern Medical School at Houston, Houston, Texas
  - The University of Texas Health Science at San Antonio, San Antonio, Texas